Online assessment and enhancement of auditory perception for speech sound errors (SCED)

Protocol NCT04858035

Document generated 10/21/2020

**PROTOCOL: STUDY 3** 

Establish the efficacy of online perceptual training for children with RSE and atypical perception

#### **OBJECTIVE:**

Evaluate whether online perceptual training improves perception and production of /r/ in children with Residual Speech Errors (RSE) who have atypical perceptual acuity, as identified by our lab-based classification norms.

## **Participants**

Sample: 10 children with RSE affecting /r/

Age range: 9;0–15;11 years, native English speakers

# Eligibility

### Residual Speech Errors (RSE):

Must have persistent speech errors specifically affecting the English rhotic /r/ sound.

## Perceptual Classification:

Must be classified as having *atypical perception* based on a laboratory-developed classification model applied to standardized perception tasks.

### Language Background:

Native speakers of English.

# • Cognitive and Language Proficiency:

Must demonstrate adequate nonverbal cognitive and language skills as assessed by standardized tests, including:

- Goldman-Fristoe Test of Articulation—Third Edition (GFTA-3): Assesses articulation of speech sounds.
- Clinical Evaluation of Language Fundamentals—Fifth Edition (CELF-5), Recalling Sentences (RS) and Formulated Sentences (FS) subtests: Evaluates expressive and receptive language functioning, focusing on sentence recall and formulation.
- o LinguiSystems Articulation Test (LAT): Measures production of specific speech sounds.

 Sentence Repetition Task (SRT): Assesses verbal memory and grammatical processing through sentence repetition.

# Hearing Screening:

Must pass an online pure-tone hearing screening at frequencies 1000 Hz, 2000 Hz, and 6000 Hz, at 30 dB intensity.

### Medical History:

Must not have a history of major neurobehavioral disorders or developmental disabilities.

#### DESIGN AND PROCEDURES

• **Design:** Multiple-baseline across-subjects design; participants randomly assigned to varying baseline durations (4–10 sessions).

#### Phases:

- o **Baseline:** Perception and production of /r/ are probed repeatedly without intervention.
- Treatment: All participants complete 12 sessions of online perceptual training (3x/week, 4 weeks).
- Maintenance: Post-treatment, perception and production are monitored for 3 sessions; no further training.

#### Assessment Measures:

### Perception:

- Online identification and category goodness judgment tasks
- For ongoing assessment, 75 items are randomly drawn (with proper balance and difficulty stratification) to avoid item memorization

#### Production:

- Standardized word probes
- Perceptual ratings are obtained from blinded online listeners

### **Perception Training (Treatment Phase)**

• **12 sessions** (30 minutes each, over 4 weeks; mostly self-administered online)

- Task 1: Focused perceptual training in a specific /r/ context with feedback; difficulty increases with improved accuracy.
- Task 2: Identification of items along a synthetic rake-wake continuum with feedback based on typical listener norms.
- Task 3: Broad perceptual training with a randomized set of items across all /r/ contexts and difficulties, with feedback.
- Clinician Monitoring: A study clinician virtually attends one session per participant each week to ensure engagement.

## **Summary Statement:**

This study will rigorously test whether online perceptual training leads to measurable improvements in both perception and production of /r/ in children with RSE and atypical perception, using a robust, randomized multiple-baseline design and blinded standardized outcome measures.